CLINICAL TRIAL: NCT03017508
Title: Double-Blind, Placebo-Controlled, Single-Dose Crossover Study Examining the Effects of Sublingual Riluzole (BHV-0223) on Public Speaking in Social Anxiety Disorder
Brief Title: Acute Anxiolytic Effects of Riluzole on Subjects With Social Anxiety Disorder
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Biohaven Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 1605017768
Record Dates: First submitted 2017-01-09; First posted 2017-01-11 (Estimated); Results first posted 2021-05-20 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-04

CONDITIONS: Social Anxiety Disorder; Performance Anxiety
Keywords: Cross-over study; Riluzole; Double-blind study; Speech task; Social Anxiety Disorder
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- BHV-0223 (Sublingual Riluzole) (Experimental): Participants will be given one dose of BHV-0223 (sublingual riluzole) 35mg before performing a 10 minute speech task. Participants will then be assessed every hour for the next three hours. There will be 2 to 10 days of washout period between the randomly assigned arms of the study.
  Interventions: Drug: BHV-0223
- Placebo (Placebo Comparator): Participants will be given one dose of an identical looking sublingual placebo before performing a 10 minute speech task. Participants will then be assessed every hour for the next three hours. There will be 2 to 10 days of washout period between the randomly assigned arms of the study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BHV-0223 — 35mg of sublingual riluzole before performing an anxiety provoking speech task. Participants will then be clinically assessed every hour for 3 hours.
  Other Names: sublingual riluzole
  Arms: BHV-0223 (Sublingual Riluzole)
Drug: Placebo — a sublingual tablet identical to the active drug will be given before performing an anxiety provoking speech task. Participants will then be clinically assessed every hour for three hours.
  Arms: Placebo

SUMMARY:
The goal of the current proposal is to examine if sublingual riluzole can reduce anxiety in people with social anxiety disorder during a public speaking task.

DETAILED DESCRIPTION:
The investigators propose conducting a double-blind, placebo controlled crossover study examining the effects of BHV-0223 on public speaking anxiety. Twenty participants with DSM-5 defined social anxiety disorder and clinically significant public speaking anxiety on the Impromptu Speech Task will be enrolled in a challenge study. Participants will be given BHV-0223 (or placebo) under double-blind crossover conditions 1 hour prior to performing each of 2 impromptu speech tasks. The two study days involving BHV-0223 (or placebo) administration and impromptu speech task will be separated by 2 to 10 days to allow for medication washout. There will be a final follow-up visit 2 to 10 days later to perform a complete Physical exam and do follow-up liver function testing and a Complete Blood Count. Our primary outcome will examine BHV-0223's effects (compared to placebo) on self-rated anxiety during the impromptu speech task. The investigators will also collect physiological measures of anxiety, clinician-rated measures of anxiety, and measures of speech performance as secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female (post-menopausal, surgically sterile, or negative pregnancy test at screening and agreement to utilize an established birth control, including complete abstinence, during the testing period) between the age of 18 and 65 yrs.
2. Meet DSM-5 criteria for social anxiety disorder by structured clinical interview (SCID) and have a LSAS public speaking subscale score >6.
3. Stable psychiatric medications. Participants must have had stable doses of all psychiatric medications for the month prior to treatment and have been on stable doses of SSRI and antidepressants for at least 1 month prior to study enrollment. As needed benzodiazepine use will be permitted as long as subjects refrain from using benzodiazepines for the 48 hours prior to the study.
4. Medically and neurologically healthy on the basis of physical examination, SMAC-20 (including LFT's, TFT's), VDRL, CBC w/ diff, urinalysis, urine toxicology, EKG, and medical history. Individuals with stable medical problems that do not have CNS effects or interfere with medications administered (e.g., oral hypoglycemics) may be included if their medications have not been adjusted in the month prior to entry;
5. Urine toxicology screen negative for drug of abuse.
6. Able to provide written informed consent according to the Yale Human Investigation Committee (HIC) guidelines.

Exclusion Criteria:

1. Positive pregnancy test
2. Breastfeeding females
3. History of substance abuse disorder (ETOH, cocaine, opiates, PCP) within the last 6 months or positive urine toxicology on screening (within the previous 6 months).
4. History of pervasive developmental disorder or psychotic disorder by DSM-IV-TR criteria.
5. Presence of dentures, braces, piercings at the time of dosing, or any physical findings in the mouth or tongue that, in the opinion of the Principal Investigator, would be likely to interfere with successful completion of the dosing procedure.
6. Participants with a medical condition that might interfere with the physiological absorption and motility (ie, gastric bypass, duodenectomy) or gastric bands.
7. Participants with any clinically significant abnormality or abnormal laboratory test results.
8. Participant has a current diagnosis of viral hepatitis (HBsAG or HVC) or a history of liver disease.
9. Participant has significant history of seizure disorder other than a single childhood febrile seizure (eg. Epilepsy)
10. Participant using any drugs known to induce or inhibit CYP 1A2 metabolism (examples of inducers: rifampin, carbamazepine, etc.; examples of inhibitors: fluvoxamine, ciprofloxacin, fluoroquinolones, etc.) within 30 days prior to the first study drug administration.
11. Participants with a history of allergic reactions to riluzole or other related drugs.
12. Participant has a history of anaphylaxis, a documented hypersensitivity reaction, or a clinically important reaction to any drug.
13. Participant has received another investigational drug or device within the 30 days (90 days for biologics) prior to the first dosing or is currently participating in an investigational study involving no drug administration.
14. Participant with clinically significant electrocardiogram (ECG) abnormalities (QTcF >450 msec) or vital sign abnormalities (systolic blood pressure lower than 90 or over 140 mmHg, diastolic blood pressure lower than 50 or over 90 mmHg, or heart rate less than 50 or over 100 bpm) at Screening or Baseline (Day -1).
15. Any reason which, in the opinion of the Principal Investigator, would prevent the participant from being in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-01; Primary Completion 2019-12 (Actual); Study Completion 2021-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael H. Bloch, MD, MS, Principal Investigator — Associate Professor
Locations (1):
- Connecticut Mental Health Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Davidson JR. Use of benzodiazepines in social anxiety disorder, generalized anxiety disorder, and posttraumatic stress disorder. J Clin Psychiatry. 2004;65 Suppl 5:29-33. PMID 15078116
- [Background] Mathew SJ, Amiel JM, Coplan JD, Fitterling HA, Sackeim HA, Gorman JM. Open-label trial of riluzole in generalized anxiety disorder. Am J Psychiatry. 2005 Dec;162(12):2379-81. doi: 10.1176/appi.ajp.162.12.2379. PMID 16330605
- [Background] Pittenger C, Coric V, Banasr M, Bloch M, Krystal JH, Sanacora G. Riluzole in the treatment of mood and anxiety disorders. CNS Drugs. 2008;22(9):761-86. doi: 10.2165/00023210-200822090-00004. PMID 18698875
- [Background] Sanacora G, Kendell SF, Levin Y, Simen AA, Fenton LR, Coric V, Krystal JH. Preliminary evidence of riluzole efficacy in antidepressant-treated patients with residual depressive symptoms. Biol Psychiatry. 2007 Mar 15;61(6):822-5. doi: 10.1016/j.biopsych.2006.08.037. Epub 2006 Dec 4. PMID 17141740
- [Background] Baker SL, Heinrichs N, Kim HJ, Hofmann SG. The liebowitz social anxiety scale as a self-report instrument: a preliminary psychometric analysis. Behav Res Ther. 2002 Jun;40(6):701-15. doi: 10.1016/s0005-7967(01)00060-2. PMID 12051488
- [Background] Ries BJ, McNeil DW, Boone ML, Turk CL, Carter LE, Heimberg RG. Assessment of contemporary social phobia verbal report instruments. Behav Res Ther. 1998 Oct;36(10):983-94. doi: 10.1016/s0005-7967(98)00078-3. PMID 9714948

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 28 participants were screened in person at the Yale Child Study Center. Of these, 22 were enrolled and 6 were excluded (2 did not have a diagnosis of Public Speaking Anxiety, 3 had a positive utox and 1 had uncontrolled hypertension).
Groups:
- Participants Randomized to BHV-0223 First and After a Washout Period of 2-10 Days Received Placebo: Participants that were randomized to receive sublingual BHV-0223 before performing a 10 minute speech task and were then followed for 3 hours. Participants were then assessed every hour for the next three hours. There was a 2 to 10 days of washout period. These participants would then receive an identical looking sublingual placebo before performing a 10 minute speech task and were followed for 3 hours.
- Participants Randomized to Placebo First and After a Washout Period of 2-10 Days Received BHV-0223: Participants that were randomized to receive sublingual placebo before performing a 10 minute speech task and were then followed for 3 hours. Participants were then assessed every hour for the next three hours. There was a 2 to 10 days of washout period. These participants would then receive sublingual BHV-0223 before performing a 10 minute speech task and were followed for 3 hours.
Period: Overall Study
Arm/Group | Participants Randomized to BHV-0223 First and After a Washout Period of 2-10 Days Received Placebo | Participants Randomized to Placebo First and After a Washout Period of 2-10 Days Received BHV-0223
Started | 12 | 10
First Intervention (1 Day) | 12 | 10
Washout (2-10 Days) | 12 | 10
Second Intervention (1 Day) | 12 | 10
Completed | 12 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Participants That Were Randomized to Receive BHV-0223 (Sublingual Riluzole) First: Participants were given one dose of BHV-0223 (sublingual riluzole) 35mg before performing a 10 minute speech task. Participants will then be assessed every hour for the next three hours. There will be 2 to 10 days of washout period between the randomly assigned arms of the study.
  BHV-0223: 35mg of sublingual riluzole before performing an anxiety provoking speech task. Participants will then be clinically assessed every hour for 3 hours.
- Participants That Were Randomized to Receive Placebo First: Participants were given one dose of an identical looking sublingual placebo before performing a 10 minute speech task. Participants will then be assessed every hour for the next three hours. There will be 2 to 10 days of washout period between the randomly assigned arms of the study.
  Placebo: a sublingual tablet identical to the active drug will be given before performing an anxiety provoking speech task. Participants will then be clinically assessed every hour for three hours.
- Total: Total of all reporting groups
Arm/Group | Participants That Were Randomized to Receive BHV-0223 (Sublingual Riluzole) First | Participants That Were Randomized to Receive Placebo First | Total
Number analyzed (Participants) | 12 | 10 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 10 | 22
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 34 [18 to 58] | 29 [20 to 40] | 31.7 [18 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 7 | 7 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 11 | 9 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 8 | 7 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 12 | 10 | 22
Visual Analogue Scale Baseline Score [Mean (Standard Deviation); unit: millimeters] — In the Visual Analogue Scale (VAS) participants are presented with a straight horizontal line of 100 mm in length and asked to mark the placement that would best describe the intensity of the anxiety felt at that moment. The left end (0mm) represents "no anxiety" and the right end (100mm) represents "the worst anxiety ever felt" by the participant.The VAS score is determined by measuring in millimeters from the left hand end of the line to the point that the patient marks, generating a numerical score along a continuum.
  millimeters | 62.25 (17.05) | 46.6 (22.5) | 55.1 (20.9)

OUTCOME MEASURES:

1. Primary Outcome: VAS-anxiety Immediately After the Impromptu Speech Task
Description: Measure Description: In the Visual Analogue Scale (VAS) participants are presented with a straight horizontal line of 100 mm in length and asked to mark the placement that would best describe the intensity of the anxiety felt at that moment. The left end (0mm) represents "no anxiety" and the right end (100mm) represents "the worst anxiety ever felt" by the participant.The VAS score is determined by measuring in millimeters from the left hand end of the line to the point that the patient marks, generating a numerical score along a continuum
Time Frame: up to 60 minutes
Measure: Mean (Standard Deviation); unit: millimeters (units on a scale)
Groups:
- BHV-0223 (Sublingual Riluzole): Participants will be given one dose of BHV-0223 (sublingual riluzole) 35mg before performing a 10 minute speech task. Participants will then be assessed immediately after finishing speech task.
  BHV-0223: 35mg of sublingual riluzole before performing an anxiety provoking speech task. Participants will then be clinically assessed immediately after finishing the speech task.
- Placebo: Participants will be given one dose of an identical looking sublingual placebo before performing a 10 minute speech task. Participants will then be assessed immediately after finishing the speech task.
  Placebo: a sublingual tablet identical to the active drug will be given before performing an anxiety provoking speech task. Participants will then be clinically assessed immediately after finishing the speech task.
Arm/Group | BHV-0223 (Sublingual Riluzole) | Placebo
Number analyzed (Participants) | 22 | 22
millimeters (units on a scale) | 54.3 (23.6) | 62.6 (13.7)
Statistical Analysis 1: Comparison: BHV-0223 (Sublingual Riluzole) vs Placebo; Paired t-test on VAS scores during speech comparing sublingual riluzole to placebo; Test type: Superiority; p = 0.056, t-test, 2 sided; Mean Difference (Final Values) = -8.34, Standard Deviation 18.34

ADVERSE EVENTS:
Time Frame: Up to 1 hour.
Arm/Group | BHV-0223 (Sublingual Riluzole) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 13/22 | 0/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BHV-0223 (Sublingual Riluzole) (N=22) | Placebo (N=22)
Temporary perioral numbing (General disorders) | 13 (13) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-28): https://cdn.clinicaltrials.gov/large-docs/08/NCT03017508/Prot_SAP_000.pdf